CLINICAL TRIAL: NCT01009515
Title: Phase II Trial of Carboplatin, Paclitaxel, and Temozolomide for Patients With Metastatic Melanoma
Brief Title: Carboplatin, Paclitaxel, and Temozolomide for Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual; target accrual not met
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0903; NCI-2011-01939 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-10-14; First posted 2009-11-06 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2015-10

CONDITIONS: Melanoma
Keywords: metastatic; melanoma; skin cancer; paclitaxel; carboplatin; temozolomide
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Skin Neoplasms | interventions — Paclitaxel; Carboplatin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy Combination (Experimental): Chemotherapy Combination of paclitaxel, carboplatin, temozolomide: Carboplatin at an AUC of 5 on Day 1, paclitaxel at 175 mg/m2 on Day 1, and temozolomide at 125 mg/m2 Day 2-Day 6, on a 28 day cycle.
  Interventions: Drug: Paclitaxel, carboplatin, temozolomide

INTERVENTIONS:
Drug: Paclitaxel, carboplatin, temozolomide — Combination chemotherapy was administered for up to 6 cycles

SUMMARY:
The number of melanoma cases has been steadily increasing over the past few decades. For many patients with metastatic melanoma, there are no effective therapies. The goal of this study is to determine whether a combination drug treatment of carboplatin, paclitaxel and temozolomide is effective in the treatment of metastatic or recurrent melanoma.

DETAILED DESCRIPTION:
Over the past several decades, significant research has been conducted to try to identify active chemotherapeutic agents for the treatment of melanoma. The rationale for combining taxanes and platinum agents is that both have activity in melanoma; in vitro and clinical data suggest synergy between these drugs when used in combination in a wide variety of tumors, including melanoma; and the toxicity profiles of these agents do not overlap. Temozolomide (a drug approved for the treatment of melanoma) has been combined with other drugs, including taxanes and platinums, in previous clinical trials for melanoma. Specifically, a previous phase I study of the combination of temozolomide, paclitaxel, and carboplatin in melanoma showed objective responses. The efficacy of this combination is now being studied in this phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients with biopsy proven advanced melanoma are eligible if there is measurable disease.
* Patients must have a life expectancy of at least 12 weeks.
* Prior surgery, immunotherapy, minimal chemotherapy (1 drug for less than 4 months), or radiotherapy for primary tumor is acceptable but must be completed at least 4 weeks from study entry, and patient should have completely recovered from such procedures.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of ≥ 1500 cells/mm3, hemoglobin > 8 g/dl, platelet count ≥ 100 000/mm3.
* Patients should have a normal hepatic function with a total bilirubin < 1.5 the upper limit of normal (ULN) and serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) < 2 times the upper limit of normal (ULN),and adequate renal function as defined by a serum creatinine ≤ 1.5 times the ULN.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and at least for 3 months.
* Patients with brain metastases are eligible if they have been appropriately treated, are asymptomatic

Exclusion Criteria:

* Pregnant women or nursing mothers are not eligible.
* Patients must not receive any other concurrent chemotherapy or radiation during this trial.
* Patients with severe medical problems that would interfere with the therapy are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2013-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Montasur Shaheen, MD, Principal Investigator — University of New Mexico
Locations (3):
- United States (3):
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - The Cancer Center at Presbyterian, Albuquerque, New Mexico

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from sites in the New Mexico Cancer Care Alliance from October, 2009 to March, 2013.
Period: Overall Study
Arm/Group | Chemotherapy Combination
Started | 19
Completed | 16
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy Combination
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White non-Hispanic | 14
  White Hispanic | 4
  Black | 1
Region of Enrollment [Number; unit: participants]
  United States | 19
Site of Metastasis [Number; unit: participants]
  Brain | 1
  Bone | 8
  Liver | 7
  Lung | 14
  Other visceral organs | 12
  Regional Lymph Nodes | 10
Previous Therapy [Number; unit: participants]
  Surgery | 16
  Radiation | 8
  Chemotherapy | 4
  Interferon | 5
  Immune Vaccines | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by physical exam and/or computerized tomography (CT): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. The Objective Response Rate (ORR) is the sum of the percentages of patients achieving CR or PR.
Time Frame: 6 months
Population: The 16 patients who completed treatment were evaluable for the endpoint of overall response rate.
Measure: Number; unit: participants
Arm/Group | Chemotherapy Combination
Number analyzed (Participants) | 16
participants
  Complete response (CR) | 1
  Partial response (PR) | 3
  Stable disease | 0
  Progressive disease (PD) | 12
  ORR (CR + PR) | 4

2. Secondary Outcome: Overall Survival
Description: The time from treatment initiation to death by any cause.
Time Frame: 2 years
Population: The 16 patients who completed treatment were evaluable for survival analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemotherapy Combination
Number analyzed (Participants) | 16
weeks | 47 [24 to 69]

3. Secondary Outcome: Safety Profile
Description: All toxicities encountered during the study by patients who receive at least one on-study treatment will be graded according to the NCI CTCAE (Version 3.0). The number of patients experiencing adverse events will be reported according to grade.
Time Frame: Up to 30 days after last on-study treatment, for up to 2 years
Population: All patients who had received at least one dose of on-study treatment were evaluable for toxicity.
Measure: Number; unit: participants
Arm/Group | Chemotherapy Combination
Number analyzed (Participants) | 19
participants
  Fatigue (Grade 1-2) | 9
  Fatigue (Grade 3-4) | 1
  Fever (Grade 1-2) | 0
  Fever (Grade 3-4) | 1
  Weight loss (Grade 1-2) | 0
  Weight loss (Grade 3-4) | 1
  Anorexia (Grade 1-2) | 1
  Anorexia (Grade 3-4) | 0
  Diarrhea (Grade 1-2) | 5
  Diarrhea (Grade 3-4) | 1
  Aspartate aminotransferase increased (Grade 1-2) | 2
  Aspartate aminotransferase increased (Grade 3-4) | 1
  Vomiting (Grade 1-2) | 2
  Vomiting (Grade 3-4) | 1
  Gastrointestinal Bleed (Grade 1-2) | 0
  Gastrointestinal Bleed (Grade 3-4) | 1
  Nausea (Grade 1-2) | 12
  Nausea (Grade 3-4) | 0
  Alanine aminotransferase increased (Grade 1-2) | 2
  Alanine aminotransferase increased (Grade 3-4) | 0
  Hyperbilirubinemia (Grade 1-2) | 1
  Hyperbilirubinemia (Grade 3-4) | 0
  Neutropenia (Grade 1-2) | 3
  Neutropenia (Grade 3-4) | 2
  Anemia (Grade 1-2) | 4
  Anemia (Grade 3-4) | 0
  Lymphopenia (Grade 1-2) | 4
  Lymphopenia (Grade 3-4) | 1
  Leukopenia (Grade 1-2) | 7
  Leukopenia (Grade 3-4) | 0
  Thrombocytopenia (Grade 1-2) | 3
  Thrombocytopenia (Grade 3-4) | 0
  Hyperglycemia (Grade 1-2) | 3
  Hyperglycemia (Grade 3-4) | 1
  Hypophosphatemia (Grade 1-2) | 0
  Hypophosphatemia (Grade 3-4) | 1
  Hypokalemia (Grade 1-2) | 3
  Hypokalemia (Grade 3-4) | 0
  Hyponatremia (Grade 1-2) | 3
  Hyponatremia (Grade 3-4) | 0
  Chest wall pain (Grade 1-2) | 1
  Chest wall pain (Grade 3-4) | 1
  Bone pain (Grade 1-2) | 2
  Bone pain (Grade 3-4) | 0
  Muscle weakness, lower limb (Grade 1-2) | 2
  Muscle weakness, lower limb (Grade 3-4) | 0
  Joint pain (Grade 1-2) | 1
  Joint pain (Grade 3-4) | 0
  Drowsiness (Grade 1-2) | 0
  Drowsiness (Grade 3-4) | 1
  Peripheral Sensory Neuropathy (Grade 1-2) | 3
  Peripheral Sensory Neutropenia (Grade 3-4) | 0
  Pericardial effusion (Grade 1-2) | 0
  Pericardial effusion (Grade 3-4) | 1
  Edema limbs (Grade 1-2) | 1
  Edema limbs (Grade 3-4) | 0
  Alopecia (Grade 1-2) | 8
  Alopecia (Grade 3-4) | 0
  Rash (Grade 1-2) | 4
  Rash (Grade 3-4) | 0
  Dry mouth (Grade 1-2) | 3
  Dry mouth (Grade 3-4) | 0

4. Secondary Outcome: Time to Progression
Description: The time from treatment initiation to disease progression or death by any cause. Progression is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by physical exam or computerized tomography (CT): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Population: The 16 patients who completed treatment were evaluable for progression-free survival.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Chemotherapy Combination
Number analyzed (Participants) | 16
weeks | 31 [19 to 58]

ADVERSE EVENTS:
Arm/Group | Chemotherapy Combination
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Combination (N=19)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Induration (Skin and subcutaneous tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy Combination (N=19)
Allergic reaction (Immune system disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hemoglobin levels decreased (Blood and lymphatic system disorders) | 4 (7)
Leukopenia (leukocytes decreased) (Blood and lymphatic system disorders) | 7 (8)
Lymphopenia (lymphocytes decreased) (Blood and lymphatic system disorders) | 5 (5)
Neutrophils decreased (Blood and lymphatic system disorders) | 3 (6)
Platelets decreased (Blood and lymphatic system disorders) | 5 (5)
Hypotension (Low blood pressure) (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (General disorders) | 3 (5)
Fatigue (General disorders) | 10 (12)
Fever (General disorders) | 1 (1)
Rigors/chills (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Alopecia (Hair loss) (Skin and subcutaneous tissue disorders) | 8 (8)
Dermatology/Skin - Other: Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Itching) (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Increased sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (2)
Anorexia (Decreased appetite) (Gastrointestinal disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Indigestion) (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 13 (24)
Taste alteration (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Edema limbs (Blood and lymphatic system disorders) | 2 (3)
Localized edema (Blood and lymphatic system disorders) | 1 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (7)
Creatinine increased (Investigations) | 3 (3)
Hyperbilirubinemia (high bilirubin levels) (Investigations) | 1 (1)
Hypercalcemia (high calcium levels) (Investigations) | 1 (1)
Hyperglycemia (high blood sugar) (Investigations) | 7 (9)
Hyperkalemia (high potassium levels) (Investigations) | 1 (1)
Hypermagnesemia (high magnesium levels) (Investigations) | 1 (1)
Hypoalbuminemia (low albumin protein levels) (Investigations) | 2 (3)
Hypocalcemia (low calcium levels) (Investigations) | 1 (1)
Hypokalemia (low potassium levels) (Investigations) | 4 (4)
Hypomagnesemia (low magnesium levels) (Investigations) | 2 (2)
Hyponatremia (low sodium levels) (Investigations) | 4 (5)
Hypophosphatemia (low phosphate levels) (Investigations) | 1 (1)
Increased lactate dehydrogenase levels (Investigations) | 4 (6)
Laboratory test abnormal (Investigations) | 1 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Depressed level of consciousness (Psychiatric disorders) | 1 (3)
Depression (Psychiatric disorders) | 2 (2)
Headache (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (5)
Ear, nose and throat examination abnormal (General disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (2)
Back pain (General disorders) | 1 (1)
Bone pain (General disorders) | 3 (6)
Buttock pain (General disorders) | 1 (1)
Chest wall pain (General disorders) | 1 (2)
Joint pain (General disorders) | 1 (3)
Neck pain (General disorders) | 1 (2)
Pain - Other (General disorders) | 3 (5)
Pain in extremity (General disorders) | 2 (2)
Pharyngolaryngeal pain (throat pain) (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Hypoxia (low blood oxygen) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Urinary frequency increased (Renal and urinary disorders) | 1 (3)
Urinary frequency decreased (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes